CLINICAL TRIAL: NCT01250990
Title: A Randomized, Double-Blind, Placebo Controlled Study Evaluating the Effects Of Niacin On Reverse Cholesterol Transport As Measured Using [1,2-3H]-Cholesterol (3H-cholesterol) in Healthy Volunteers.
Brief Title: Effect of Niacin on Transport of HDL and Relationship to Atherogenic Lipoproteins and Lipolysis
Acronym: ENTHRALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Richard Dunbar, Research Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 811956; K23HL091130 (NIH)
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Dyslipidemias
Keywords: Niacin; HDL; Reverse cholesterol transport
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niacin (Active Comparator): Niacin taken orally for 12 weeks at the highest tolerated dose (up to 6 grams), and at least 2 grams daily and up to the maximum approved dose. Subjects will initiate therapy with Niaspan and will advance to Niacor as tolerated.
  Interventions: Drug: Niacin
- Placebo (Placebo Comparator): Placebo tablet with 50 mg niacin for the first 4 weeks to maintain blinding of the study team and subjects, changed to pure placebo after that.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Niacin — Niacin taken orally for 12 weeks at the highest tolerated dose (up to 6 grams), and at least 2 grams daily and up to the maximum approved dose. Subjects will initiate therapy with Niaspan and will advance to Niacor as tolerated.
  Other Names: Niacor and Niaspan
  Arms: Niacin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study looks at whether niacin improves reverse cholesterol transport (RCT) in healthy volunteers. 3H-Cholesterol will be used to measure RCT by analyzing changes in the tracer activity in total plasma, lipoproteins, red blood cells (RBCs) and stool. The hypothesis is that niacin augments reverse cholesterol transport.

DETAILED DESCRIPTION:
The study will use 3H-cholesterol bound to albumin (particulate cholesterol) to assess the ability of high density lipoprotein (HDL) to transport cholesterol to the liver to be eliminated. This process is called Reverse Cholesterol transport and is one of the main mechanisms by which HDL protect against atherosclerotic cardiovascular disease. The availability of a method to assess RCT is important for the development of new drugs which affect RCT and may result in useful treatments for atherosclerosis.

This study will evaluate the use of radiolabeled particulate cholesterol administered intravenously in association with albumin, as a method to study reverse cholesterol transport (RCT) in humans before and after treatment by niacin by analyzing changes in the tracer activity in total plasma and lipoproteins. The study population is healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 75 inclusive
* HDL cholesterol >= 25 mg/dL in all subjects, and <= 60 mg/dL in men and <= 70 mg/dL in women
* Women must be of non-childbearing potential. They must have been surgically sterilized at least 6 months prior to screening or be postmenopausal. Postmenopausal women must have no regular menstrual bleeding for at least 2 years prior to inclusion.
* Subjects must be in good overall health.
* Subjects must be able to comprehend and willing to provide a signed Institutional Regulatory Board (IRB) approved Informed Consent Form.
* Subjects must be willing to comply with all study-related procedures.
* Subjects must weigh at least 140 pounds to participate in the HDL kinetics Substudy.

Exclusion Criteria:

* Clinically-manifest cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease
* History of diabetes mellitus or fasting glucose > 126 mg/dL at the screening visit
* Presence of New York Heart Association (NYHA) Class III or IV chronic heart failure or unstable angina pectoris
* History of any other endocrine disease
* History of a non-skin malignancy within the previous 5 years
* Anemia defined as hemoglobin less than 12 g/dL
* Renal insufficiency as defined by creatinine ³ 1.3 mg/dl
* Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition
* Uncontrolled hypertension (Systolic >160 mm Hg and/or Diastolic >100 mmHg on two consecutive measurements
* Use of warfarin, or any known coagulopathy and /or elevated Prothrombin time/Partial Thromboplastin Time (PT/PTT) >1.5 x upper limit of normal (ULN)
* Self-reported history of Human immunodeficiency virus (HIV) positive
* Previous organ transplantation
* Clinical evidence of liver disease or liver injury as indicated by abnormal liver function tests such as Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2x ULN, or self-reported history of positive for Hepatitis B or Hepatitis C
* Any major surgical procedure that occurred within the previous 3 months of the screening visit
* History of illicit drug abuse (< 1 year)
* Regular use of alcoholic beverages (> 2 drinks/day)
* Body mass index (BMI) > 35 kg/m2 or < 18.5 kg/m2
* Administration of an investigational drug within 6 weeks prior to the screening visit
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study will be excluded.
* Use of daily lipid-altering therapy prior to the initiation of study medication is exclusionary under the following circumstances (washout of non-statins is permitted):

  * Statins within 4 weeks
  * Niacin > 250 mg/ day within 6 weeks: Advicor, Niaspan, Niacor, Simcor, Slo-Niacin, or supplemental niacin
  * Fibrates within 12 weeks: fenofibrate (Antara, Lofibra, Tricor, Triglide), gemfibrozil (Lopid), or clofibrate
  * Enterically active lipid-altering drugs within 4 weeks: colestipol (Colestid), cholestyramine (Questran), colesevelam (Welchol), ezetimibe (Zetia, Vytorin), orlistat (Xenical, Alli)
  * Red yeast rice
  * Fish oil > 2 g/day within 4 weeks: Lovaza (née Omacor), numerous supplements
  * Altered dose of a selective estrogen receptor modulator (SERM) within 4 weeks
* History of severe intolerance of niacin
* Men who plan to conceive a child within 3 months of the conclusion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Dunbar, MD MSTR, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niacin | Placebo
Started | 11 | 11
Completed | 7 | 9
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Rate of Appearance of 3H Cholesterol in the Total HDL Fraction Before and After 12 Weeks of Treatment With Niacin
Description: Subjects were injected with a bolus of 3-H cholesterol mixed with human serum albumin as an intravenous bolus. This injected labelled cholesterol is taken up by macrophages. The rate of appearance of labelled cholesterol in plasma HDL- cholesterol is a measure of reverse cholesterol transport. We assessed HDL cholesterol enrichment as percent of injected tritiated tracer appearing in plasma total HDL cholesterol between 60 and 240 minutes post-injection expressed as percent 3-H cholesterol/mol HDL cholesterol/hour. The tracer study was performed at baseline and after 12 weeks of niacin or placebo.
Time Frame: Baseline and 12 weeks
Population: Of the 22 subjects enrolled, only subjects who completed the baseline and 12 week reverse cholesterol transport studies were included in the final outcome analysis.
Measure: Mean (95% Confidence Interval); unit: %/mol/h
Arm/Group | Niacin | Placebo
Number analyzed (Participants) | 7 | 9
%/mol/h
  Pre-treatment | 3.24 [2.22 to 4.26] | 4.16 [3.20 to 5.12]
  Post-treatment | 2.61 [1.59 to 3.63] | 3.72 [2.76 to 4.67]
Statistical Analysis 1: Comparison: Niacin vs Placebo; This is a pilot study to assess the effects of niacin on reverse cholesterol transport. The null hypothesis is that niacin has no effect on reverse cholesterol transport; Test type: Superiority or Other; p = 0.8, t-test, 2 sided — p value is for comparison between changes in reverse cholesterol transport in niacin versus placebo groups after 12 weeks of treatment

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Niacin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes